CLINICAL TRIAL: NCT03689855
Title: Ramucirumab and Atezolizumab After Progression on Any Immune Checkpoint Blocker in NSCLC (RamAtezo-1)
Brief Title: Ramucirumab and Atezolizumab After Progression on Any Immune Checkpoint Blocker in NSCLC
Acronym: RamAtezo-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201810163
Record Dates: First submitted 2018-09-27; First posted 2018-10-01 (Actual); Results first posted 2022-08-11 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Non-small Cell Lung Cancer; Non Small Cell Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ramucirumab; atezolizumab; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ramucirumab + Atezolizumab (Experimental): * Ramucirumab will be given intravenously over the course of an hour on an outpatient basis on Day 1 of each 21-day cycle at a dose of 10 mg/kg.
  * Atezolizumab will be given intravenously on an outpatient basis on Day 1 of each 21-day cycle at a dose of 1200 mg.
  Interventions: Drug: Ramucirumab; Drug: Atezolizumab; Procedure: Peripheral blood draw; Procedure: Biopsy

INTERVENTIONS:
Drug: Ramucirumab — Ramucirumab is an investigational agent for this trial and will be supplied by Lilly Oncology, free of charge to the patient.
  Other Names: Cyramza
Drug: Atezolizumab — The initial dose will be administered over 60 minutes (+/- 15 minutes). If the first infusion is tolerated without infusion-associated events, the second infusion may be delivered over 30 minutes (+/- 10 minutes).
  Other Names: Tecentriq
Procedure: Peripheral blood draw — -Baseline and Cycle 2 Day 1
Procedure: Biopsy — * If archival biopsy tissue not available, participant will undergo biopsy at baseline
  * When feasible, a repeated tumor biopsy will be obtained between Cycles 2 and 3 after the scheduled CT scan.

SUMMARY:
Data suggests that combining ramucirumab with immunotherapy in non-small cell lung cancer (NSCLC) patients who have previously received immune checkpoint blockers (ICBs) may be more effective than traditional therapy. The investigators propose a pilot study to test the combination of ramucirumab and atezolizumab in patients with advanced-stage NSCLC patients previously treated with ICB.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed squamous or non-squamous non-small cell lung cancer. Patients with known EGFR or ALK mutations are eligible only if they have received at least one line of targeted therapy for these mutations.
* Availability of archival biopsy tissue or willingness to undergo a "baseline" biopsy prior to initiation of the trial for biomarker analysis, including PD-L1 by IHC. Note: Results of PD-L1 testing are not required for enrollment.
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan, as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam.
* Prior use of an immune checkpoint blocker alone or in combination therapy.
* At least 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/cumm
  * Platelets ≥ 100,000/cumm
  * Hemoglobin ≥ 9.0 g/dL
  * Total bilirubin ≤ 1.5 x ULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x ULN or 5.0 x ULN in the setting of liver metastasis
  * Serum creatinine ≤ 1.5 x ULN or CrCl ≥ 40 mL/min. if serum creatinine is >1.5 times the ULN, a 24-hour urine collection to calculate creatinine clearance must be performed
* Adequate coagulation function as defined by:

  * INR ≤ 1.5
  * PTT/aPTT < 1.5 x ULN
* Note: Patients on full-dose anticoagulation must be on a stable dose (minimum duration 14 days) of oral anticoagulant or low molecular weight heparin (LMWH). If receiving warfarin, the patient must have an INR ≤3.0. For heparin and LMWH there should be no active bleeding (that is, no bleeding within 14 days prior to first dose of protocol therapy) or pathological condition present that carries a high risk of bleeding (for example, tumor involving major vessels or known varices).
* Urinary protein ≤ 1+ on dipstick or routine urinalysis; if urine dipstick or routine analysis is ≥ 2+, a 24-hour urine collection for protein must demonstrate < 1000 mg of protein in 24 hours to allow participation
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Treatment with cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to Cycle 1, Day 1.

  *Note: Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea or premedication for contrast dye allergy) are eligible. The use of inhaled corticosteroids for chronic obstructive pulmonary disease (COPD) and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.
* A history of other malignancy ≤ 3 years previous with the exception of patients with a negligible risk of metastasis or death and with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, or ductal carcinoma in situ treated surgically with curative intent) or undergoing active surveillance per SOC management (e.g., Rai Stage 0 chronic lymphocytic leukemia, prostate cancer with Gleason score ≤ 6 and prostate-specific antigen (PSA ≤ 10 ng/mL, etc.).
* Currently receiving any other investigational agents.
* Symptomatic or untreated asymptomatic brain metastases. Patients with treated brain metastases are eligible if they are clinically stable with regard to neurologic function, off steroids after cranial irradiation (whole brain radiation therapy, focal radiation therapy, and stereotactic radiosurgery) ending at least 2 weeks prior to randomization, or after surgical resection performed at least 28 days prior to randomization. The patient may have no evidence of Grade ≥1 CNS hemorrhage based on pretreatment MRI or IV contrast CT scan (performed within 21 days before randomization).
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to atezolizumab, ramucirumab, any other immune checkpoint blockade, chimeric or humanized antibodies, fusion proteins, or other agents used in the study.
* Receiving chronic antiplatelet therapy, including aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs, including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents. Once-daily aspirin use (maximum dose 325 mg/day) is permitted.
* Arterial or venous thromboembolic event, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to enrollment.
* Uncontrolled or poorly controlled hypertension (> 160 mmHg systolic or > 100 mmHg diastolic for > 4 weeks) despite standard medical management.
* Gastrointestinal perforation, and/or fistula, or risk factors for perforation within 6 months prior to enrollment.
* Grade 3 or 4 gastrointestinal bleeding within 3 months prior to enrollment.
* History of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis.

  *Note: Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone are eligible. Patients with controlled type 1 diabetes mellitus on a stable insulin regimen are eligible.
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug-induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest CT scan.
* Hemoptysis (defined as bright red blood or ≥ ½ teaspoon) within 2 months prior to Cycle 1 Day 1 or with radiographic evidence of intratumor cavitation or radiologically documented evidence of major blood vessel invasion or encasement by cancer.
* Serious or non-healing would, ulcer, or bone fracture within 28 days prior to Cycle 1 Day 1.
* Undergone major surgery within 28 days prior to Cycle 1 Day 1, or minor surgery/subcutaneous venous access device placement within 7 days prior to Cycle 1 Day 1, or has elective or planned major surgery to be performed during the course of the clinical trial.
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, cirrhosis at a level of Child-Pug B or worse, cirrhosis (any degree) with a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis (defined as ascites from cirrhosis requiring diuretics or paracentesis), fatty liver, and inherited liver disease.

  --Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection (defined as, HBV surface antigen (HBsAg) positive and HBV core antibody (HbcAb) positive with reflex positive HBV DNA. Note: Patients with past or resolved hepatitis B infection (defined as having a negative HBsAg test and a positive HBcAb test or treated HCV with negative HCV RNA are eligible.
* Known HIV-positivity.
* Active tuberculosis.
* Administration of a live, attenuated influenza vaccine within 4 weeks before Cycle 1 Day 1 or at any time during the study.
* Severe infections within 2 weeks prior to Cycle 1 Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia. Received oral or intravenous (IV) antibiotics within 2 weeks prior to Cycle 1 Day 1. Note: Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible.
* History of deep venous thrombosis, pulmonary embolism, or any other significant thromboembolism (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant") during the 3 months prior to Cycle 1 Day 1.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test within 7 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2024-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Morgensztern, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xing P, Wang M, Zhao J, Zhong W, Chi Y, Xu Z, Li J. Study protocol: A single-arm, multicenter, phase II trial of camrelizumab plus apatinib for advanced nonsquamous NSCLC previously treated with first-line immunotherapy. Thorac Cancer. 2021 Oct;12(20):2825-2828. doi: 10.1111/1759-7714.14113. Epub 2021 Aug 18. PMID 34409776
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ramucirumab + Atezolizumab
Started | 21
Completed | 17
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ramucirumab + Atezolizumab
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 67 [42 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: * ORR: percentage of participants with a complete or partial response
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: At 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ramucirumab + Atezolizumab
Number analyzed (Participants) | 21
Participants | 1

2. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: * CBR is defined as the percentage of patients who have achieved responses (complete or partial) or stable disease.
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: At 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ramucirumab + Atezolizumab
Number analyzed (Participants) | 21
Participants | 16

3. Secondary Outcome: Toxicity and Tolerability as Measured by Number of Participants Who Experienced Adverse Events
Description: -Measured by NCI-CTCAE version 5.0.
Time Frame: Through 30 days after completion of treatment (estimated to be 4 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Ramucirumab + Atezolizumab
Number analyzed (Participants) | 21
Participants
  Grade 1-2 anemia | 8
  Grade 3-5 atrial fibrillation | 1
  Grade 3-5 pericardial effusion | 1
  Grade 1-2 ear pain | 1
  Grade 1-2 hypothyroidism | 4
  Grade 1-2 eye pain | 1
  Grade 1-2 abdominal pain | 1
  Grade 3-5 ascites | 1
  Grade 1-2 colitis | 1
  Grade 1-2 constipation | 5
  Grade 1-2 diarrhea | 6
  Grade 1-2 dyspepsia | 1
  Grade 1-2 dysphagia | 2
  Grade 1-2 mucositis oral | 1
  Grade 1-2 nausea | 10
  Grade 1-2 oral pain | 1
  Grade 1-2 stomach pain | 1
  Grade 1-2 vomiting | 7
  Grade 1-2 non-cardiac chest pain | 1
  Grade 1-2 chills | 4
  Grade 1-2 edema limbs | 3
  Grade 1-2 infusion related reaction | 1
  Grade 1-2 vascular access complication | 1
  Grade 1-2 alanine aminotransferase increased | 3
  Grade 1-2 alkaline phosphatase | 4
  Grade 1-2 aspartate aminotransferase increased | 1
  Grade 1-2 creatinine increased | 4
  Grade 1-2 hemoglobin increased | 2
  Grade 1-2 lipase increased | 1
  Grade 1-2 lymphocyte count decreased | 5
  Grade 1-2 neutrophil count decreased | 3
  Grade 1-2 platelet count decreased | 4
  Grade 1-2 serum amylase increased | 3
  Grade 1-2 thyroid stimulating hormone increased | 7
  Grade 1-2 weight loss | 5
  Grade 3-5 weight loss | 1
  Grade 1-2 white blood cell decreased | 3
  Grade 1-2 anorexia | 8
  Grade 3-5 anorexia | 1
  Grade 1-2 dehydration | 1
  Grade 1-2 hypercalcemia | 1
  Grade 1-2 hyperglycemia | 3
  Grade 1-2 hyperkalemia | 2
  Grade 1-2 hypoalbuminemia | 6
  Grade 1-2 hypocalcemia | 4
  Grade 1-2 hypoglycemia | 2
  Grade 1-2 hyponatremia | 6
  Grade 3-5 hyponatremia | 1
  Grade 1-2 hernia right groin | 1
  Grade 1-2 pain right groin | 1
  Grade 1-2 rib pain | 1
  Grade 1-2 arthralgia | 3
  Grade 1-2 flank pain | 1
  Grade 1-2 generalized muscle weakness | 2
  Grade 1-2 myalgia | 5
  Grade 1-2 neck pain | 1
  Grade 1-2 osteonecrosis of jaw | 1
  Grade 3-5 pain in extremity | 1
  Grade 3-5 bilateral vocal cord paralysis | 1
  Grade 3-5 right vocal fold paralysis | 1
  Grade 1-2 cognitive disturbance | 2
  Grade 1-2 dizziness | 3
  Grade 1-2 dysgeusia | 2
  Grade 1-2 dysphasia | 1
  Grade 1-2 headache | 9
  Grade 1-2 memory impairment | 1
  Grade 1-2 peripheral motor neuropathy | 1
  Grade 1-2 peripheral sensory neuropathy | 1
  Grade 1-2 somnolence | 1
  Grade 3-5 somnolence | 1
  Grade 1-2 stroke | 1
  Grade 1-2 transient ischemic attacks | 1
  Grade 1-2 anxiety | 1
  Grade 1-2 confusion | 1
  Grade 1-2 delirium | 1
  Grade 1-2 insomnia | 2
  Grade 1-2 hematuria | 4
  Grade 1-2 proteinuria | 12
  Grade 1 pelvic pain | 1
  Grade 1-2 hemoptysis | 1
  Grade 1-2 allergic rhinitis | 3
  Grade 3-5 atelectasis | 1
  Grade 1-2 cough | 8
  Grade 1-2 dyspnea | 3
  Grade 3-5 dyspnea | 1
  Grade 1-2 epistaxis | 2
  Grade 1-2 hiccups | 1
  Grade 1-2 nasal congestion | 1
  Grade 1-2 oropharyngeal pain | 1
  Grade 1-2 sore throat | 2
  Grade 1-2 alopecia | 1
  Grade 1-2 hyperhidrosis | 1
  Grade 1-2 rash maculo-papular | 1
  Grade 1-2 hypertension | 15
  Grade 3-5 hypertension | 3
  Grade 1-2 hypotension | 3

4. Secondary Outcome: Overall Survival (OS)
Time Frame: Through 2 years after completion of treatment (median length of follow-up 16.3 months, full range=2.3-45.6 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab + Atezolizumab
Number analyzed (Participants) | 21
months | 16.3 [7.1 to 20.9]

5. Secondary Outcome: Progression-free Survival (PFS)
Description: -PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Time Frame: Through 2 years after completion of treatment (median length of follow-up 16.3 months, full range=2.3-45.6 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab + Atezolizumab
Number analyzed (Participants) | 21
months | 1.0 [1.0 to 2.3]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment through 30 days after the last administration of the study treatment. All-cause mortality was collected from start of treatment until completion of follow-up. The median length of treatment was 92 days (full range 49 days-812 days). The median length of follow-up was 16.3 months (full range 2.3 months-45.6 months).
Arm/Group | Ramucirumab + Atezolizumab
All-Cause Mortality (participants affected / at risk) | 15/21
Serious Adverse Events (participants affected / at risk) | 10/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ramucirumab + Atezolizumab (N=21)
Atrial fibrillation (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Portal hypertension (Hepatobiliary disorders) | 1
COVID-19 (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 1
Stroke (Nervous system disorders) | 1
Transient ischemic attacks (Nervous system disorders) | 1
Vocal cord paralysis (Nervous system disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ramucirumab + Atezolizumab (N=21)
Anemia (Blood and lymphatic system disorders) | 9
Ear pain (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 4
Eye pain (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 10
Oral pain (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Chills (General disorders) | 4
Edema limbs (General disorders) | 3
Fatigue (General disorders) | 9
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 2
Conjunctivitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Thrush (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Vulval infection (Infections and infestations) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 1
Creatinine increased (Investigations) | 4
Hemoglobin increased (Investigations) | 2
Lipase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 4
Serum amylase increased (Investigations) | 3
Thyroid stimulating hormone increased (Investigations) | 7
Weight loss (Investigations) | 6
White blood cell decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 9
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Hernia right groin (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pain right groin (Musculoskeletal and connective tissue disorders) | 1
Rib pain (Musculoskeletal and connective tissue disorders) | 1
Cognitive disturbance (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 2
Dysphasia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 8
Memory impairment (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Right vocal fold paralysis (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Hematuria (Renal and urinary disorders) | 4
Proteinuria (Renal and urinary disorders) | 12
Pelvic pain (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 17
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/55/NCT03689855/Prot_SAP_000.pdf